CLINICAL TRIAL: NCT03519958
Title: An Observational, Multi-centre Study on EGFR T790M Mutation Testing Practices and Outcomes Conducted Among Locally Advanced/Metastatic NSCLC Patients Who Progressed on Previous EGFR Tyrosine-kinase Inhibitor (TKI) Therapy in Hong Kong
Brief Title: Epidermal Growth Factor Receptor (EGFR) T790M Mutation Testing Practices in Hong Kong
Status: Withdrawn | Type: Observational
Why Stopped: The study direction does not longer aligns the sponsor's strategy
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00019
Record Dates: First submitted 2018-02-19; First posted 2018-05-09 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma for T7909M ctDNA testing Urine for T7909M ctDNA testing Tissue (optional)

GROUPS / COHORTS (1):
- EGFR NSCLC Progressed on EGFR TKI: Patients with EGFR NSCLC who have progressed following EGFR TKI therapy will undergo plasma-tissue testing
  Interventions: Diagnostic Test: Plasma-tissue testing

INTERVENTIONS:
Diagnostic Test: Plasma-tissue testing — EGFR T790M mutation plasma-tissue testing in NSCLC patients who progressed on previous EGFR TKI

SUMMARY:
To describe the T790M mutation status of patients with locally advanced/metastatic NSCLC who progressed on previous EGFR TKI treatment in a real-world setting.

DETAILED DESCRIPTION:
This is a multi-center, observational study of patients with locally advanced/metastatic NSCLC who progressed on previous EGFR TKI treatment. Eligible patients will be recruited from participating sites in Hong Kong over a 12 months enrolment period.

Plasma and urine samples will be collected from enrolled patients. Plasma circulating tumor DNA (ctDNA) and urine ctDNA will be analyzed by droplet digital PCR (ddPCR) for detection of T790M mutation and EGFR sensitizing mutations. Patients who are T790M plasma-negative, regardless of the urine testing results, will be recommended to undergo re-biopsy (defined as tissue sampling or cytology sampling), tissue/cytology T790M testing, and to provide a second plasma sample for a second plasma T790M test (tested by ddPCR).

Enrolled patients who subsequently receive osimertinib treatment will be followed up as per routine practice at the investigational site. Patient data will be collected for 12 months or until death or loss to follow-up, whichever occurs earlier, from the first prescription of osimertinib. All clinical decisions will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria

* Provision of written informed consent
* Locally advanced (stage IIIB) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy
* Confirmed EGFR sensitizing mutation (exon 19 deletion or exon 21 L858R ) in medical record
* Progressed on previous EGFR TKI treatment, based on physician judgement, with or without additional lines of treatment
* Suggested to undergo T790M mutation testing by treating physician, based on physician judgement

Exclusion Criteria

* Had been treated with osimertinib or any other 3rd generation T790M inhibitors
* Enrollment in studies that prohibit participation in this observational study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol locally advanced or metastatic NSCLC patients with confirmed EGFR sensitizing mutation, who progressed after EGFR TKI treatment (i.e.,gefitinib, erlotinib, afatinib), and are suggested to undergo T790M mutation testing by their treating physicians in participating sites in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
EGFR T790M mutation prevalance | 3 years
  Based on the plasma-tissue testing algorithm in NSCLC patients who progressed on previous EGFR TKI therapy

SECONDARY OUTCOMES:
Proportion of Valid Tissue T790M Testing Result | 3 years
  Proportion of study subjects who have a valid tissue/cytology T790M testing result after receiving a negative plasma test result for the T790M mutation
T790M Plasma Outcome | 3 years
  Proportions of study subjects who are T790M plasma-negative
False Negative Proportation | 3 years
  Proportion of study subjects who are T790M plasma-negative but T790M tissue/cytology-positive
Reasons for not performing re-biopsy | 3 years
  reasons given for not performing re-biopsy and tissue/cytology testing after obtaining a negative plasma test result
Demographics | Baseline
  Demographics of T790M-positive subjects and T790M-negative subjects
Disease Characteristics | 3 years
  Disease characteristics of T790M-positive subjects and T790M-negative subjects
Number of particapants with complications assoicated with re-biopsy | 3 years
  Number of particapants with complications assoicated with tissue/cytology re-biopsy
Clinical Outcomes in T790M plasma-positive subejects | 3 years
  Clinical outcomes after osimertinib treatment between study subjects who are T790M plasma-positive
Clinical Outcomes in urine-positive | 3 years
  Clinical outcomes after osimertinib treatment between study subjects who are urine-positive
Clinical Outcomes in tissue/cytology-positive | 3 years
  Clinical outcomes after osimertinib treatment between study subjects who are tissue/cytology-positive

OTHER OUTCOMES:
Concordance | 3 years
  To analyze the concordance of T790M mutation status as determined by urine, plasma, and tissue/cytology T790M testing

CONTACTS AND LOCATIONS:
Overall Officials: James Ho, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong